CLINICAL TRIAL: NCT06294821
Title: 4-Aminopyridine to Delay Carpal Tunnel Release or Resolve Carpal Tunnel Syndrome
Brief Title: 4AP for Carpal Tunnel Syndrome (CTS)
Acronym: CTS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Elfar (Other)
Responsible Party: Sponsor-Investigator, John Elfar, Tenured Professor, Chairman, Department of Orthopaedic Surgery, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00003845
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Compression Neuropathy; Carpal Tunnel Syndrome
Keywords: 4 aminopyridine; carpal tunnel syndrome; CTR; 4AP; CTS; Carpal tunnel release; compression neuropathy
MeSH Terms: conditions — Tomaculous neuropathy; Carpal Tunnel Syndrome | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4-aminopyridine (Active Comparator): Study drug: dalfampridine (generic) 10mg ER capsule
  Interventions: Drug: 4-Aminopyridine
- Placebo (Placebo Comparator): Placebo-1 capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 4-Aminopyridine — Subjects will receive either the active study drug (4-aminopyridine) or placebo to determine the effects of 4AP on carpal tunnel syndrome
  Other Names: 4AP
  Arms: 4-aminopyridine
Other: Placebo — Subjects will receive either the active study drug (4-aminopyridine) or placebo to determine the effects of 4AP on carpal tunnel syndrome
  Arms: Placebo

SUMMARY:
The investigators have found recent promising data supporting the use of a currently FDA approved drug, 4-aminopyridine, in the treatment of nerve injury including compression neuropathy. The purpose of this research is determine whether 4-aminopyridine can treat carpal tunnel syndrome or delay the need for formal surgical release in patients with known carpal tunnel syndrome who would otherwise undergo surgery.

DETAILED DESCRIPTION:
Carpal tunnel syndrome affects somewhere between 3 and 10% of the Unites States population. Symptoms associated with this disorder include numbness and tingling in the radial three digits of the hand. These symptoms often cause sleeplessness. They have been attributed to work related activities. The diagnosis of carpal tunnel syndrome is made clinically. Several confirmatory tests exist in the setting of carpal tunnel syndrome. In the United States the gold standard diagnostic for carpal tunnel syndrome is electrodiagnostic evaluation. This notwithstanding, recent literature suggests that other diagnostic methods including ultrasound evaluation of the median nerve at the carpal tunnel as well as clinical diagnostic criteria are sufficient to adequately and specifically diagnose carpal tunnel syndrome.

Several treatments exist for carpal tunnel syndrome. Treatment range from non-operative braces or positional movements. Moving on to intervention treatments there are several injections that have been used to treat carpal tunnel syndrome. Carpal Tunnel Syndrome is most definitively and completely treated by surgical release of the median nerve at the carpal tunnel. Surgical releases themselves have been performed under a variety of techniques from formal median nerve exploration to mini-open release as well endoscopic release. Resolution of symptoms after carpal tunnel release has been regarded as the gold standard to which other treatments can be compared.

Several registries of compression neuropathy patients have been compiled. These registries reveal that non-invasive assessment with standardize validated questionnaires can be used to measure the progression of symptomology, and the resolution of treatment. Given the history and wealth of experience in the diagnosis and treatment in this condition, it's natural to ask are there non-operative pharmacological treatments that may delay or remove the need for carpal tunnel release surgery. Certainly, the comparison to surgical decompression as the gold standard is desirable.

More research is needed to evaluate the role of 4-aminopyridine (4AP) in the treatment of compression neuropathy. The investigational treatment will be used to test the hypothesis that 4AP improves symptoms and electrodiagnostic parameters in carpal tunnel syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with non-traumatic carpal tunnel syndrome without any other confounding diagnosis (e.g. cubital tunnel syndrome, cervical nerve compression)
* Standard of care EDX testing within 6 months of study enrollment
* Cognitive ability to report sensory and motor deficit during examination.
* Able to complete twice daily dosing of 4-AP for the entire 6 week treatment period.
* Adults subject aged 18-90
* Ability to give written informed consent.
* Capable of safely undergoing electrodiagnostic testing (EDX).
* Availability for all study visits.

Exclusion Criteria:

* Inability to complete twice daily dosing during 6 week treatment period.
* History of multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of hypersensitivity to AMPYRA® or 4-aminopyridine
* Current use of aminopyridine medications, including other compounded 4-AP
* Suspected renal impairment based on the Choyke questionnaire.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Results of symptomatic improvement in the Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ) | Baseline (prior to study treatment) to 56 weeks post treatment
  Improvement of Carpal Tunnel Syndrome symptoms will be measured using the Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ) - a validated patient reported outcome measure. The scale contains 6 items on the severity and frequency of night and daytime numbness, tingling and pain. Each item is scored on a 5-point Likert scale from 1 (no symptoms) to 5 (most severe symptoms). Subjects will complete a baseline questionnaire prior to treatment initiation. The questionnaire will be completed all study visit following initiation of treatment until the final study visit at 56 weeks post treatment.
Results of symptomatic improvement in the Michigan Hand Outcomes Questionnaire (MHQ) | Baseline (prior to study treatment) to 56 weeks post treatment.
  Improvement of Carpal Tunnel Syndrome symptoms will be measured with standardized validated outcomes measure, the Michigan Hand Outcomes Questionnaire (MHQ) for improvement in carpal tunnel symptomatology. The MHQ is a tool used to assess patients with hand disorders through the measurement of 6 health domains: overall hand function, activities of daily living, pain, work performance, aesthetics, and patient satisfaction. In the pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance. Baseline measures will be completed prior to treatment and repeated at each study visit with the final outcome questionnaire completed at the final, 56 week visit.

SECONDARY OUTCOMES:
Electrodiagnostic improvement following treatment | Baseline (prior to study treatment) and 8 weeks post treatment.
  Nerve conduction velocity improvement > 10% compared to pre-treatment nerve conduction velocity. Electrodiagnostic studies will be completed as part of standard of care prior to initiation of treatment and repeated at 8 weeks post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Elfar, MD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No